CLINICAL TRIAL: NCT04359342
Title: Effects of High-intensity Interval Training Combined With Post-exercise Protein Supplementation on Cardiorespiratory Fitness in Untrained Individuals: a Double-blind Placebo-controlled Trial
Brief Title: Protein Supplementation and HIIT: Impact on Cardiorespiratory Fitness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-HIIT Study
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Primary Prevention; Health Promotion
Keywords: Aerobic exercise; Cardiorespiratory Fitness; High-intensity interval training (HIIT); Resistance training; Protein intake
MeSH Terms: interventions — Proteins; Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Parallel Assignment parallel-group, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomized, double-blind placebo-controlled study. Participants and Outcome Assessors will not be aware of the arm to which the participants are allocated (double-blinded masking).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIIT + protein (Experimental): High-intensity interval training (HIIT) combined with protein supplementation
  Interventions: Dietary Supplement: HIIT + protein
- HIIT + placebo (Placebo Comparator): High-intensity interval training (HIIT) combined with placebo
  Interventions: Dietary Supplement: HIIT + placebo
- HIIT and resistance training + protein (Experimental): High-intensity interval training (HIIT) and resistance training combined with protein supplementation
  Interventions: Dietary Supplement: HIIT and resistance training + protein
- HIIT and resistance training + placebo (Placebo Comparator): High-intensity interval training (HIIT) and resistance training combined with placebo
  Interventions: Dietary Supplement: HIIT and resistance training + placebo

INTERVENTIONS:
Dietary Supplement: HIIT + protein — 8-week supervised exercise program consisting of high-intensity interval training (HIIT).
  HIIT: 10x1 min at 85-95% HRmax divided by low intensity recovery periods. Three exercise sessions per week. Participants receive 40 g of a commercially available protein supplement administered as a shake after every exercise session.
  Arms: HIIT + protein
Dietary Supplement: HIIT + placebo — 8-week supervised exercise program consisting of high-intensity interval training (HIIT).
  HIIT: 10x1 min at 85-95% HRmax divided by low intensity recovery periods. Three exercise sessions per week. Participants receive 40 g of a commercially available iso-caloric placebo (Maltodextrin) administered as a shake after every exercise session.
  Arms: HIIT + placebo
Dietary Supplement: HIIT and resistance training + protein — 8-week supervised exercise program consisting of high-intensity interval training (HIIT) and resistance training (RST).
  HIIT: 5x1 min at 85-95% HRmax divided by low intensity recovery periods. RST: 3-set resistance training using weight machines to train all major muscle groups with an individual intensity corresponding to 70-80% of one repetition maximum. Two exercise sessions per week. Participants receive 40 g of a commercially available protein supplement administered as a shake after every exercise session.
  Arms: HIIT and resistance training + protein
Dietary Supplement: HIIT and resistance training + placebo — 8-week supervised exercise program consisting of high-intensity interval training (HIIT) and resistance training (RST).
  HIIT: 5x1 min at 85-95% HRmax divided by low intensity recovery periods. RST: 3-set resistance training using weight machines to train all major muscle groups with an individual intensity corresponding to 70-80% of one repetition maximum. Two exercise sessions per week. Participants receive 40 g of a commercially available iso-caloric placebo (Maltodextrin) administered as a shake after every exercise session.
  Arms: HIIT and resistance training + placebo

SUMMARY:
The aim of this study is to investigate the effects of an 8-week high-intensity interval training (HIIT) or HIIT plus resistance training program combined with post-exercise protein supplementation on cardiorespiratory fitness and cardiometabolic risk indices in previously untrained individuals.

ELIGIBILITY:
Inclusion Criteria:

• Sedentary Lifestyle over at least 6 months prior to the study

Exclusion Criteria:

* Pregnancy, Lactation
* Psychological disorders, epilepsy, sever neurological disorders
* Participation in other exercise- or nutrition studies within the last 6 months
* coronary heart disease, heart failure
* malignant disease
* severe rheumatic or neurological disease
* severe/unstable hypertension (resting RR: >180/>110 mmHg)
* severely restricted lung function (FEV1 <60%)
* unstable Diabetes mellitus
* severe orthopedic disease/restriction
* acute / chronic infectious diseases
* Electronic implants (defibrillator, pacemaker)
* Persons in mental hospitals by order of authorities or jurisdiction

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness (CRF) | 8 weeks
  CRF will be assessed by measuring maximum oxygen uptake (VO2max)
Muscle strength (only in groups with resistance training) | 8 weeks
  Maximum strength (Fmax) of the major muscle groups (chest, upper back, lower back, abdominals and legs) will be estimated through submaximal tests, based on the performance of multiple repetitions.

SECONDARY OUTCOMES:
Cardiometabolic Risk Score (MetS-Z-Score) | 8 weeks
  MetS-Z-Score will be calculated from each individual's measures of waist circumference (cm), mean arterial blood pressure (mmHg), Glucose (mg/dL), triglycerides (mg/dL), and HDL-cholesterol (mg/dL), based on equations specific to sex.
Muscle mass | 8 weeks
  Muscle mass (kg) will be measured by Bioelectrical Impedance Analysis (BIA)
Fat mass | 8 weeks
  Fat mass (kg) will be measured by Bioelectrical Impedance Analysis (BIA)
Insulin sensitivity | 8 weeks
  Insulin sensitivity will be estimated using homeostasis model assessment index (HOMA)
Inflammation status | 8 weeks
  Inflammation status will be assessed by measuring blood levels (mg/L) of c-reactive protein (CRP) and high-sensitivity c-reactive protein (hs-CRP)
Health-related quality of life | 8 weeks
  Health-related quality of life will be assessed by using the standardized and validated EQ-5D-5L Questionnaire, consisting of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The patient ticks the box next to the most appropriate statement in each dimension (scale: 1-5; lower value = better outcome). The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.The EQ VAS records the patient's self-rated health on a vertical visual analogue scale (0-100, higher value = better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Reljic, Dr., Principal Investigator — University Erlangen Nuremberg Medical School; Yurdagül Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany